CLINICAL TRIAL: NCT02894463
Title: Uncontrolled Prospective Single-center Study Aimed at Detecting Potential Abuse of Nitrous Oxide in Children During Dental Care
Brief Title: Study Aimed at Detecting Potential Abuse of Nitrous Oxide in Children During Dental Care
Acronym: MEOPAeDent
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC14_0213
Record Dates: First submitted 2016-08-11; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-08

CONDITIONS: Periodontal Disease
Keywords: dental care; emeno; abuse
MeSH Terms: conditions — Periodontal Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: questionnaire

SUMMARY:
The aim of this study is to evaluate the potential risk of abusive behavior for children in care using nitrous oxide for dental care.

DETAILED DESCRIPTION:
The expected prospects are therefore maintaining surveillance around the MEOPA following his release from hospital reserves, but also to ensure that the MEOPA not an addictive potential in the context of its use in dentistry. The results of this study will in any case to secure its application for dental care.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 15 years
* Requiring dental care under MEOPA
* Not opposing, as well as his parents, his participation in the study
* Not having difficulties tracking (going on holiday, imminent change, remoteness, lack of motivation)

Exclusion Criteria:

Excluded patients are those whose dental care can be made to the vigil state, or on the contrary, will present a number of important care, justifying general anesthesia.

Also excluded will be children whose parents no longer have parental authority or whose parents are divorced or divorcing.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients seen in consultation EMENO and being younger than 15 years will be offered this study.
  This is a population of non-cooperative patients to dental care or with a disability limiting their cooperation.
  A quick questionnaire will be submitted in the consultations EMENO the SSC, the children after their parents' permission.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
presence of clear signs that the child is trying to extend the contact MEOPA ( questionnaire ) | Baseline
  hand gesture to keep the mask over the nose and / or mouth, verbalization of the desire to keep the mask over the nose and / or mouth, to extend the negotiation contac

CONTACTS AND LOCATIONS:
Overall Officials: Tony Prud'homme, Dr, Principal Investigator — Nantes University Hospital